CLINICAL TRIAL: NCT05660564
Title: Aswan University Hospital
Brief Title: Preputial Graft Urethroplasty in Primary Repair of Hypospadias
Acronym: Hypospadias
Status: Completed | Type: Observational
Sponsor: Sarah Magdy Abdelmohsen (Other)
Collaborators: Aswan University Hospital (Other)
Responsible Party: Sponsor-Investigator, Sarah Magdy Abdelmohsen, Lecturer, Aswan University Hospital
Organization: Aswan University Hospital (Other)
Other Study IDs: AswanUH5
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Completed

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: DIGU Dorsal inlay preputial graft urethroplasty — Using a scalpel, a midline incision is made from the meatus to the end of the plate .
  The edge of the distal glans should not be incised to avoid meatal stenosis. The depth of this relaxing incision depends on the plate's width and depth, but in all cases, it extends down to the corpora cavernosa. Degloving of the penile skin to the penoscrotal junction If a minimal chord is present, it should be corrected.
  From the inner prepuce, a free graft was measured, harvested, defatted, and stitched to the UP. With interrupted 6/0 polyglactin sutures running from the old meatus to the tip of the glans, the graft was secured to the medial edges of the incised plate. Depending on the location of the meatus, the characteristics of the UP, and the depth of the midline incision, the graft width and length varied in each case.

SUMMARY:
Introduction: Hypospadias repair is debated. There has been no perfect procedure until this moment. A graft is sometimes needed to fundamentally strengthen the narrow urethral plate.

Patients and methods: The study included a child who had primary distal or mid-penile hypospadias at the age of 6 months or more, a urethral plate less than 8 mm in a non-circumcised penis, and was operated on using the Snodgraft technique.

DETAILED DESCRIPTION:
Patients and methods This study was designed as a prospective cross-sectional study during the period from May 2018 to October 2019. The study included hypospadias patients who were admitted to a hypospadias clinic at a university hospital.

Inclusion criteria were that a child complained of primary distal or mid-penile hypospadias at age 6 months or more, had a urethral plate less than 8 mm, and had a non-circumcised penis. Children with redo hypospadias, significant Chordee (30 percent or more), non-preservable plates, circumcised patients, and proximal hypospadias were excluded.

History has been taken from the parent of the patient in the form of the direction of the urine stream, manifestation of urinary tract infection, past history and previous repair, family history of hypospadias among first-degree relatives, history of hormonal intake (local or systemic), gestational history as a history of acute or chronic diseases, and exposure to drugs or environmental endocrinological disrupters.

Physical examination as body weight, other associated congenital anomalies, and other medical problems. Local examination of the external genitalia includes the penile size and length (normal or small penis). The meatus was examined for its position, caliber, and presence or absence of surrounding shiny skin. The prepuce was examined for shape and width (complete or incomplete). The shape and width of the glens were examined (cleft, incomplete cleft, flat). The urethral plate was examined for its width, length, or associated urethral dysplasia. If and to what extent there is or is not penile curvature, scrotal transposition, or penile rotation, Examination of the scrotal wall is either well developed or underdeveloped. Examination of the scrotal contents: palpation of the testis, whether it is present or absent (undescended), its site, size, bilateral symmetry, or any associated problem such as a congenital hernia or hydrocele.

Routine investigations such as CBCS, PT, PC, urine analysis, and urine culture if necessary. Abdominopelvic ultrasonography to rule out associated congenital anomalies. Before general anesthesia was administered, all patients received a preoperative dose of IV 3rd generation cephalosporins (50 mg/kg). Then the caudal block was done to reduce the post-operative pain. Patients are placed in a supine position, and sterilization and toweling are done to expose the external genitalia.

Preoperative measurements were taken after induction of anesthesia before the start of the operation; penile girth, urethral plate length, urethral plate width, vertical length of the glans (Fig. 2A), and maximum width of the glans .

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were that a child complained of primary distal or mid-penile hypospadias at age 6 months or more, had a urethral plate less than 8 mm, and had a non-circumcised penis.

Exclusion Criteria:

* . Children with redo hypospadias, significant Chordee (30 percent or more), non-preservable plates, circumcised patients, and proximal hypospadias were excluded.

Ages: 6 Months to 8 Years | Sex: All
Age Groups: Child
Study Population: The study included hypospadias patients who were admitted to a hypospadias clinic at a university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
75% success rate | one and half year

CONTACTS AND LOCATIONS:
Locations (1):
- Sarah Magdy Abdelmohsen, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol